CLINICAL TRIAL: NCT03267212
Title: Acute Effect of Ventilatory Support During Exercise in Spinal Cord Injury
Acronym: NIV-Ex-CS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, J. Andrew Taylor, Principle Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SpauldingRH-2
Record Dates: First submitted 2017-08-22; First posted 2017-08-30 (Actual); Results first posted 2020-03-30 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-03

CONDITIONS: Spinal Cord Injury
Keywords: Functional Electrical Stimulation (FES)-Rowing; Ventilatory support
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators and technicians helping for performing the test and encouraging the patient will be blind. Only one investigator will monitor the ventilation during the test and won't be blind but won't be participating to any encouragement or data acquisition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Non-invasive Ventilation(NIV) (Active Comparator): Subjects will perform FES-row testing while receiving bi-level positive airway pressure ventilation applied through a full face-mask.
  Interventions: Device: Non-invasive ventilation(NIV); Other: Functional Electrical Stimulation Row Training (FESRT)
- Sham Non-invasive ventilation(NIV) (Sham Comparator): Subjects will perform FES-row testing while receiving sham ventilation applied through a full face-mask.
  Interventions: Device: Sham Non-invasive ventilation(NIV); Other: Functional Electrical Stimulation Row Training (FESRT)

INTERVENTIONS:
Device: Non-invasive ventilation(NIV) — The ventilator will be set in spontaneous mode with a ramp to reach a minimal pressure of 12 centimeters of water (cmH2O) during inspiration and 3 cmH2O during expiration.
  Arms: Non-invasive Ventilation(NIV)
Device: Sham Non-invasive ventilation(NIV) — The ventilator will be set in spontaneous mode with a ramp to reach a maximal pressure of 5 centimeters of water (cmH2O) during inspiration and 3 cmH2O during expiration.
  Arms: Sham Non-invasive ventilation(NIV)
Other: Functional Electrical Stimulation Row Training (FESRT) — FESRT couples volitional arm and electrically controlled leg exercise to allow whole body exercise training

SUMMARY:
The investigators have an existing exercise program (N>70) with a unique population of individuals with spinal cord injury (SCI) who have been enrolled in Functional Electrical Stimulation - Rowing Training (FES-RT) for at least 6 months. Previous data in the laboratory from this exercise platform has recently showed that respiratory restriction in SCI reduces inspiratory capacity in direct relation to lesion level, and those with high level injuries have the greatest compromise. As a result, the increase in ventilatory requirements with FES training results in an imbalance between ventilatory capacity and greater whole body skeletal muscle demand after FES rowing training. Hence, external ventilatory support could improve the ability to exercise train and hence enhance the adaptations to chronic exercise in high level SCI. If our hypothesis is correct, this indicates that maximal aerobic capacity in these individuals exceeds maximal voluntary ventilation. It will be important to determine however the consistency of this response and at what level of injury it is not observed. In parallel of the study # NCT02865343, the investigators will recruit here a population of subjects who have completed six months of FES-row exercise training across a range of SCI level (C5-T12). Hence, the investigators will be able to determine the consistency of the effect and the dependence of the effect on SCI level. Some of them with level >T3 may also enroll in training effect study with NIV or sham NIV (NCT02865343))

DETAILED DESCRIPTION:
Regular aerobic exercise with sufficient intensity can improve overall health, however daily energy expenditure is low in those with SCI, especially in those with high level lesions. The investigators have developed Functional Electrical Stimulation Row Training (FESRT) that couples volitional arm and electrically controlled leg exercise, increasing the active muscle and resulting in benefits of large muscle mass exercise. Despite the potential for enhancing aerobic capacity, those with high level lesions (C4 to T2) have a remaining obstacle to attaining higher work capacities. They have the greatest pulmonary muscle denervation and our preliminary work suggests this limits the aerobic capacity that can be achieved with FESRT. External ventilatory support could improve the ability to reach higher level of peak ventilation and hence enhance the ability to exercise in high level SCI. Therefore, the investigators hypothesize that the use of NIV during FESRT will reduce ventilatory limits to exercise, leading to increased aerobic capacity in high level SCI. The aims are to examine the acute effect of NIV on FES-row VO2max in subjects with both high and low level SCI. The investigators have access to a large (N>70) and unique population of individuals with SCI who have been enrolled in FESRT for at least 6 months. Roughly half have SCI between C4 and T2 and half with lower injury levels (<T3). 15 individuals who have FES row trained for at least 6 months will perform FES-VO2max row tests on separate days with and without the use of NIV to determine maximal aerobic capacity and ventilation. Both FES-VO2max Row tests will be performed at least 48-hours apart. Both tests will be performed with the NIV set-up but with and without use of the NIV support in a random order. The level of inspiratory pressure will be individually set during a familiarization test. The investigators will assess maximal aerobic capacity, minute ventilation, tidal volume and cardiac output during FES-rowing. Based on current data, it is hypothesized that only those with higher level of injury (> T3) will experience further increases in aerobic capacity when using the NIV support. This exploratory/developmental research project will determine feasibility and effectiveness of this approach to exercise and will lay the groundwork for a larger, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 to 70 (IRB amendment to change maximal age from 60 to 70 years old approved on 9/20/17)
* Have had SCI (at neurological level C5-T12 with American Spinal Injury Association grade A or B or C)
* Medically stable
* Have FES-row trained for >6 months

Exclusion Criteria:

* Hypertension(Blood pressure>140/90 mmHg)
* Significant arrhythmias
* Coronary disease
* Chronic respiratory disease
* Diabetes
* Renal disease
* Cancer
* Epilepsy
* Current use of cardioactive medications
* Current grade 2 or greater pressure ulcers at relevant contact sites
* Other neurological disease
* Peripheral nerve compression or rotator cuff tears that limit the ability to row
* History of bleeding disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Andrew Taylor, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Hospital Cambridge, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vivodtzev I, Picard G, Cepeda FX, Taylor JA. Acute Ventilatory Support During Whole-Body Hybrid Rowing in Patients With High-Level Spinal Cord Injury: A Randomized Controlled Crossover Trial. Chest. 2020 May;157(5):1230-1240. doi: 10.1016/j.chest.2019.10.044. Epub 2019 Nov 16. PMID 31738927

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-invasive Ventilation First, Then Sham Ventilation: All subjects performed FES-row testing while receiving bi-level positive airway pressure ventilation first and then Sham ventilation applied through a full face-mask.
  Non-invasive ventilation(NIV): The ventilator was set in spontaneous mode with a ramp to reach a minimal pressure of 12 centimeters of water (cmH2O) during inspiration and 3 cmH2O during expiration.
  Sham Non-invasive ventilation(NIV): The ventilator was set in spontaneous mode with a ramp to reach a maximal pressure of 5 centimeters of water (cmH2O) during inspiration and 3 cmH2O during expiration.
  Functional Electrical Stimulation Row Training (FESRT): FESRT couples volitional arm and electrically controlled leg exercise to allow whole body exercise training
- Sham Ventilation First, Then Non-invasive Ventilation: All subjects performed FES-row testing while receiving Sham bi-level positive airway pressure ventilation first and then true ventilation applied through a full face-mask.
  Non-invasive ventilation(NIV): The ventilator was set in spontaneous mode with a ramp to reach a minimal pressure of 12 centimeters of water (cmH2O) during inspiration and 3 cmH2O during expiration.
  Sham Non-invasive ventilation(NIV): The ventilator was set in spontaneous mode with a ramp to reach a maximal pressure of 5 centimeters of water (cmH2O) during inspiration and 3 cmH2O during expiration.
  Functional Electrical Stimulation Row Training (FESRT): FESRT couples volitional arm and electrically controlled leg exercise to allow whole body exercise training
Period: First Intervention
Arm/Group | Non-invasive Ventilation First, Then Sham Ventilation | Sham Ventilation First, Then Non-invasive Ventilation
Started | 6 (Non-invasive ventilation) | 9 ("First Intervention (1 day)", "Washout (2 days)", and "Second Intervention (1 day)")
High SCI | 2 | 5
Low SCI | 4 | 4
Completed | 5 | 6
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1
Period: Washout (Min 2 Days / Max 7 Days)
Arm/Group | Non-invasive Ventilation First, Then Sham Ventilation | Sham Ventilation First, Then Non-invasive Ventilation
Started | 5 | 6
Completed | 4 | 6
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Second Intervention
Arm/Group | Non-invasive Ventilation First, Then Sham Ventilation | Sham Ventilation First, Then Non-invasive Ventilation
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Fifteen participants with SCI of American Spinal Injury Association Grade A or B or C, aged 40 (21 - 70) years and with a BMI of 27.2 kg/m2 (18-37). All participants were Not Hispanic or Latino but one participant had an unknown ethnicity. All participants were white but one participant was Black or African American.
Groups:
- Non-invasive Ventilation(NIV) vs. Sham Ventilation: All subjects performed FES-row testing while receiving bi-level positive airway pressure ventilation (or Sham ventilation) applied through a full face-mask. The tests were performed in a random order.
  Non-invasive ventilation(NIV): The ventilator was set in spontaneous mode with a ramp to reach a minimal pressure of 12 centimeters of water (cmH2O) during inspiration and 3 cmH2O during expiration.
  Sham Non-invasive ventilation(NIV): The ventilator was set in spontaneous mode with a ramp to reach a maximal pressure of 5 centimeters of water (cmH2O) during inspiration and 3 cmH2O during expiration.
  Functional Electrical Stimulation Row Training (FESRT): FESRT couples volitional arm and electrically controlled leg exercise to allow whole body exercise training
Arm/Group | Non-invasive Ventilation(NIV) vs. Sham Ventilation
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 40 [21 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
Body Mass Index [Mean (Full Range); unit: Kg/m2] | 27 [18 to 37]

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Aerobic Capacity During FES-row Testing
Description: Volunteers performed 2 separate maximal FES-row tests, one with Non-invasive Ventilation Support and one with Sham-NIV
Time Frame: Day 0 and Day 2
Population: 10 subjects completed both NIV and Sham tests
Measure: Mean (Standard Deviation); unit: L/min
Groups:
- Non-invasive Ventilation: Volunteers performed a maximal FES-row tests with Non-invasive Ventilation Support
- Sham Ventilation: Volunteers performed a maximal FES-row tests with Sham-NIV
Arm/Group | Non-invasive Ventilation | Sham Ventilation
Number analyzed (Participants) | 10 | 10
L/min | 1.83 (0.76) | 1.82 (0.64)

2. Secondary Outcome: Change in Cardiac Output During FES-row Testing
Description: Volunteers performed 2 separate maximal FES-row tests, one with Non-invasive Ventilation Support and one with Sham-NIV
Time Frame: Day 0 and Day 2
Population: Due to technical issues, only one participant could perform both tests (NIV and sham) for this outcome
Measure: Number; unit: L/min
Arm/Group | Non-invasive Ventilation | Sham Ventilation
Number analyzed (Participants) | 1 | 1
L/min | 9.6 | 10.3

3. Secondary Outcome: Change in Minute Ventilation During FES-row Testing
Description: Volunteers performed 2 separate maximal FES-row tests, one with Non-invasive Ventilation Support and one with Sham-NIV
Time Frame: Day 0 and Day 2
Population: Participants who completed both NIV and sham tests
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Non-invasive Ventilation | Sham Ventilation
Number analyzed (Participants) | 10 | 10
L/min | 38.8 (9.6) | 40.3 (10.0)

4. Secondary Outcome: Change in Tidal Volume During FES-row Testing
Description: Volunteers performed 2 separate maximal FES-row tests, one with Non-invasive Ventilation Support and one with Sham-NIV
Time Frame: Day 0 and Day 2
Population: Participants who completed both NIV and sham tests
Measure: Mean (Standard Error); unit: L
Arm/Group | Non-invasive Ventilation | Sham Ventilation
Number analyzed (Participants) | 10 | 10
L | 1.6 (0.3) | 1.4 (0.3)

ADVERSE EVENTS:
Time Frame: 20 months
Description: This study was investigating the effect of an additional tool to help respiratory function during a single session of exercise. Adverse events has been collected during the whole period of the study.
Arm/Group | Non-invasive Ventilation | Sham Ventilation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
The repeatability of maximal incremental exercise tests is difficult in Spinal cord injury, increasing the variability of the measure. Higher number of participants will be necessary to study the effect of NIV on the aerobic capacity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT03267212/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT03267212/ICF_001.pdf